CLINICAL TRIAL: NCT01433926
Title: Observational, Cross-sectional Study to Analyze the Characteristics of Disseminated Her2+ Breast Cancer Patients Treated With Trastuzumab That Have Reached Complete Remission, Partial Remission or Stabilization of Disease During More Than 3 Years
Brief Title: Characteristics of Disseminated Her2+ Breast Cancer Patients Treated With Trastuzumab That Have Reached Complete, Partial Remission or Stabilization of Disease During More Than 3 Years
Acronym: LongHer
Status: Completed | Type: Observational
Sponsor: Asociación para el Progreso de la Oncología en Málaga (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: LongHer
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: HER-2 Positive Breast Cancer
Keywords: Breast cancer.; Trastuzumab.; Complete remission.
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — primary tumor, preserved in paraffin
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Main objective: To analyze the clinical and biological characteristics of patients with disseminated breast cancer HER2 + treated with trastuzumab that have achieved a complete remission, partial or stable disease for a period exceeding 3 years.

In addition, there will be a sub-genetic analysis of patients in whom there is availability a sample of primary tumor preserved in paraffin. This sub-analysis will not interfere with routine clinical practice, as the tumor samples based on which will be held on genetic profile, have been preserved in paraffin was extracted from the primary tumor to the patient.

DETAILED DESCRIPTION:
SECONDARY OBJECTIVES:

* To determine the frequency of patients achieving partial response or stable disease for a period exceeding 3 years.
* Know the time to complete or partial remission or to achieve stabilization of the disease.
* Know the length of the complete or partial remission or time to disease stabilization of patients.
* Knowing the pattern of treatment that has achieved complete or partial remission or stabilization of disease and duration.
* Knowledge of overall survival.
* Knowing the toxicity of prolonged administration of trastuzumab.
* Identify the primary tumor genes HER-2 associated with such prolonged responses.

The source document will be in all cases the clinical history and in the case of patients selected for the sub-genetic analysis, the report resulting from it.

The study is carried out by filling a notebook of electronic data collection that gathers all available information contained in medical records.

The sub-genetic analysis will be performed at the Hospital de la Paz. Both, the processing of samples and conducting the analysis using qRT-PCR, will be performed in this hospital.

All data are stored, ensuring the confidentiality, security and authenticity .The forms must be reviewed by the monitor.

Once recorded the data, the database will be revised and monitored to submit those records in which there are inconsistencies or missing information . Following the closure of the database will be a report which will present the results of the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

1. Women older than 18.
2. Patients with disseminated breast cancer with overexpression of HER-2 (IHC 3 + or FISH +).
3. Patients who have been treated with trastuzumab (Herceptin ®).
4. Complete remission, partial or stable disease for a period exceeding 3 years, except for exclusive cerebral progression.
5. Patients who have given their written informed consent.

Exclusion Criteria:

1- Patients with remission achieved with surgery or less than three months of treatment with trastuzumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with disseminated breast cancer, HER-2 3+ or FISH+.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Alba, Study Chair — Hospital Virgen de la Victoria
Locations (39):
- Spain (39):
  - Hospital oncológico de Galicia, A Coruña, A Coruña
  - Hospital de Alcoy Virgen de los Lirios, Alcoy, Alicante
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Pau, Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital de Igualada, Igualada, Barcelona
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital General Yagüe, Burgos, Burgos
  - Hospital San Pedro de Alcántara, Cáceres, Cáceres
  - Hospital Punta de Europa, Algeciras, Cádiz
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Clínico San Cecilio, Granada, Granada
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital de Guadalajara, Guadalajara, Guadalajara
  - Hospital de Donostia, San Sebastián, Guipúzcoa
  - Hospital Juan Ramón Jiménez, Huelva, Huelva
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital de Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - MD Anderson, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hsopital Doce de Octubre, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Quirón, Pozuelo de Alarcón, Madrid
  - Hospital Virgen de la Victoria, Málaga, Málaga
  - Hospital Serranía de Ronda, Ronda, Málaga
  - Hospital Central Universitario de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Nuestra Señora De Valme, Seville, Sevilla
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital La Fe, Valencia, Valencia
  - Hospital Río Hortega, Valladolid, Valladolid
  - Hospital Provincial de Zamora, Zamora, Zamora
  - Hospital Miguel Servet, Zaragoza, Zaragoza